CLINICAL TRIAL: NCT05042388
Title: Mindful MAT Adherence: Mindfulness-Based Relapse Prevention (MBRP) to Improve Extended-release Naltrexone (XR-NTX) Adherence and Drug-use Outcomes for Opioid Use Disorder (OUD)
Brief Title: Mindfulness-Based Relapse Prevention to Improve Medication Assisted Treatment Adherence and Drug-use Outcomes for Opioid Use Disorder
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: West Chester University of Pennsylvania (Other)
Collaborators: National Institute on Drug Abuse (NIDA) (NIH)
Responsible Party: Principal Investigator, Michael Gawrysiak, Associate Professor of Psychology, West Chester University of Pennsylvania
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: R15DA050102 (NIH); 1R15DA050102-01A1 (NIH)
Record Dates: First submitted 2021-08-27; First posted 2021-09-13 (Actual); Last update posted 2024-12-19 (Actual); Status verified 2024-12

CONDITIONS: Opioid-use Disorder
Keywords: Addiction; Relapse Prevention; Opioid; Mindfulness
MeSH Terms: conditions — Opioid-Related Disorders; Behavior, Addictive

STUDY DESIGN:
Intervention Model Description: Participants will be randomly assigned to 1 of 2 conditions: MBRP+TAU or TAU.
Who Masked: Outcomes Assessor
Masking Description: The assessor collecting information from the participants during each post-discharge follow-up phase will be blind to which treatment condition the participant was assigned to.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Mindfulness-Based Relapse Prevention - Rolling Admission (MBRP-RA) (Experimental): Group intervention comprised of didactics and trainings in cognitive behavioral therapy relapse prevention skills and mindfulness meditation.
  Interventions: Behavioral: Mindfulness-Based Relapse Prevention - Rolling Admission (MBRP-RA)
- Treatment-As-Usual (TAU) (Active Comparator): Standard procedure for residential treatment program. Includes: supportive group therapy; Narcotics Anonymous/12-Step Programming; music, art, and animal therapy; psycho-education on issues related to mental health and substance use disorders; and medication counseling. No aspect of the treatment-as-usual services provided entails mindfulness training or components of mindfulness training.
  Interventions: Behavioral: Treatment-As-Usual

INTERVENTIONS:
Behavioral: Mindfulness-Based Relapse Prevention - Rolling Admission (MBRP-RA) — Integrates evidenced-based practices to decrease the probability and severity of relapse for those in addiction recovery. MBRP incorporates components from CBT relapse prevention and includes training in meditation practices as a means to foster increased awareness of emotional and cognitive experiences. MBRP also includes training in brief informal meditations aimed at increasing awareness and adaptive response to drug cues and negative affect.
  Arms: Mindfulness-Based Relapse Prevention - Rolling Admission (MBRP-RA)
Behavioral: Treatment-As-Usual — Standard treatment programming procedures for all individuals residing within the residential treatment program. Includes: supportive group therapy; Narcotics Anonymous/12-Step Programming; music, art, and animal therapy; psycho-education on general issues related to mental health and SUDs; and medication counseling.
  Arms: Treatment-As-Usual (TAU)

SUMMARY:
This proposal aims to determine whether an adjunctive Mindfulness-Based Relapse Prevention (MBRP) treatment program improves Medication Assisted Treatment (MAT) adherence and reduces drug-use among opioid use disorder (OUD) patients. The broad long-term objectives of this project are to investigate how integrative pharmacological and behavioral treatments improve OUD treatment outcomes. Participants for this study will include 200 patients diagnosed with opioid use disorder (OUD), that are enrolled in a 60-day residential addiction treatment program and prescribed MAT for OUD. Participants will be randomly assigned to a MBRP behavioral treatment condition or a non-MBRP treatment-as-usual (TAU) control condition as part of their treatment within the residential addiction treatment program. All participants will be monitored for three-months following their discharge from the program to test the hypotheses that MBRP participants, relative to TAU participants, will (1) demonstrate greater MAT adherence following discharge, and (2) evidence reduced drug-use following discharge.

DETAILED DESCRIPTION:
Medically detoxified OUD patients enrolling into a 60-day residential program will be randomized to either MAT Treatment-As-Usual (TAU; n=100) or TAU+MBRP (MBRP; n=100) as part of their residential treatment and followed for 3-months post-discharge to assess MAT adherence and drug-use. All participants (n=200) will participate in residential TAU (i.e., MAT, supportive group therapy), will be scheduled monthly MAT appointments per discharge treatment procedures, and will complete assessments at baseline, post- treatment, and 1-, 2-, and 3-month follow-ups. Study Aims include:

AIM 1 (PRIMARY): Compare impact of TAU versus TAU+MBRP on medication adherence and drug-use outcomes. Hypotheses: Relative to TAU, TAU+MBRP participants will demonstrate a) greater MAT adherence measured at follow-up timepoints, and b) reduced drug-use (i.e., self-report, urine drug-screens [UDS]) measured at discharge and follow-up timepoints. AIM 2: Determine whether the beneficial effects of TAU+MBRP on outcome are mediated by improvements in opioid craving and dispositional mindfulness. Hypotheses: TAU+MBRP participants will report greater improvements in distress tolerance and mindfulness, relative to TAU, which will mediate treatment outcomes (i.e., MAT adherence, reduced drug use and positive-UDS). EXPLORATORY AIM 3: Determine effects of baseline factors on treatment outcomes. Hypotheses: More severe trauma exposure (i.e., increased number of traumas) and greater posttraumatic stress symptom severity will result in poorer treatment adherence (i.e., reduced MAT follow-up appointments) and worse drug-use outcomes (i.e., increased self-reported drug use, positive-urine drug-screens) throughout each the follow-up assessments among TAU participants but not among MBRP participants.

Study Design Overview: In an randomized controlled trial design, patients enrolling into a residential addiction treatment center will be randomized to TAU (i.e., MAT, supportive group therapy) or TAU+MBRP with comparisons being made between MBRP (n=100) and treatment-as-usual (TAU; n=100) on assessment measures collected at baseline, prior to residential discharge, and at 1, 2, and 3-month follow-up time points. To address AIM 1 (TAU+MBRP, Adherence and Drug-Use): participants will be randomly assigned to receive TAU or MBRP+TAU, during their residence within an inpatient treatment setting and will complete assessments at enrollment, prior to discharge, and at 1, 2, and 3-months follow-up to assess MAT adherence and drug-use. Comparisons, on assessment measures collected at follow-up, will be made between treatment conditions to determine if MBRP+TAU results in greater number MAT adherence, fewer positive UDS, reduced drug-craving, and increased mindfulness. AIM 2 (MBRP Mechanisms of Change): Will determine whether the beneficial effects of MBRP on treatment outcome (i.e., MAT adherence, drug-use) are mediated by increases in mindfulness and distress tolerance. AIM 3 (Predictors of MAT Adherence): will examine the extent to which prior trauma-exposure and PTSD symptom severity moderates MAT adherence and drug-use outcomes, among TAU participants (but not MBRP participants), following discharge from residential treatment.

ELIGIBILITY:
Inclusion Criteria:

1. An informed consent document voluntarily signed and dated by the subject.
2. Subject must understand and be able to read and write in English.
3. Enrollment in residential treatment at study site.
4. Physically healthy males and females, aged 18 or older, who meet criteria for opioid use disorder (based on Diagnostic and Statistical Manual 5th Edition criteria) as their primary diagnosis, who are enrolled in residential treatment at the collaborating study site.
5. Subject must be willing to be randomized to treatment condition.
6. Subjects who are willing and able to comply with scheduled visits and other study procedures.

Exclusion Criteria:

1. Meets current or lifetime DSM-V criteria for schizophrenia or any psychotic disorder or organic mental disorder, including dementia-related psychosis as determined by the semi-structured interview.
2. Presence of any other psychiatric disorder that in the opinion of the PI will interfere with completion of the study or place the patient at heightened risk through participation in the study.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 105 (Actual)
Dates: Start 2021-08-01 (Actual); Primary Completion 2024-08-20 (Actual); Study Completion 2024-08-20 (Actual)

PRIMARY OUTCOMES:
Adherence to Medication Assisted Treatment (MAT) | Assessed 1 month following discharge from residential addiction treatment facility (approximately 30 days post-discharge).
  Whether participant receives MAT during post-residential-treatment discharge follow-up phase
Adherence to Medication Assisted Treatment (MAT) | Assessed 2 months following discharge from residential addiction treatment facility (approximately 60 days post-discharge).
  Whether participant receives MAT during post-residential-treatment discharge follow-up phase
Adherence to Medication Assisted Treatment (MAT) | Assessed 3 months following discharge from residential addiction treatment facility (approximately 90 days post-discharge).
  Whether participant receives MAT during post-residential-treatment discharge follow-up phase
Drug Use (Urine Drug Screens) | Assessed 1 month following discharge from residential addiction treatment facility (approximately 30 days post-discharge).
  Assessed via medical record review of urine drug-screens (when possible)
Drug Use (Urine Drug Screens) | Assessed 2 months following discharge from residential addiction treatment facility (approximately 60 days post-discharge)
  Assessed via medical record review of urine drug-screens (when possible)
Drug Use (Urine Drug Screens) | Assessed 3 months following discharge from residential addiction treatment facility (approximately 90 days post-discharge)
  Assessed via medical record review of urine drug-screens (when possible)
Drug Use (self-report) | Assessed 1 month following discharge from residential addiction treatment facility (approximately 30 days post-discharge).
  Assessed via participant completion of research-assistant administered time-line followback interview (follow-up phone call)
Drug Use (self-report) | Assessed 2 months following discharge from residential addiction treatment facility (approximately 60 days post-discharge).
  Assessed via participant completion of research-assistant administered time-line followback interview (follow-up phone call)
Drug Use (self-report) | Assessed 3 months following discharge from residential addiction treatment facility (approximately 90 days post-discharge).
  Assessed via participant completion of research-assistant administered time-line followback interview (follow-up phone call)
Opioid Craving | Assessed immediately prior to discharge from residential addiction treatment facility (approximately 50 days post-admission).
  Opioid craving will be assessed using the Opioid Craving Scale (McHugh et al., 2014). Scores for this scale range from 0 to 30, with higher scores reflecting greater craving for opioids (i.e., worse outcome).
Opioid Craving | Assessed 1 month following discharge from residential addiction treatment facility (approximately 30 days post-discharge).
  Opioid craving will be assessed using the Opioid Craving Scale (McHugh et al., 2014). Scores for this scale range from 0 to 30, with higher scores reflecting greater craving for opioids (i.e., worse outcome).
Opioid Craving | Assessed 2 month following discharge from residential addiction treatment facility (approximately 60 days post-discharge).
  Opioid craving will be assessed using the Opioid Craving Scale (McHugh et al., 2014). Scores for this scale range from 0 to 30, with higher scores reflecting greater craving for opioids (i.e., worse outcome).
Opioid Craving | Assessed 3 month following discharge from residential addiction treatment facility (approximately 90 days post-discharge).
  Opioid craving will be assessed using the Opioid Craving Scale (McHugh et al., 2014). Scores for this scale range from 0 to 30, with higher scores reflecting greater craving for opioids (i.e., worse outcome).

SECONDARY OUTCOMES:
Dispositional Mindfulness | Assessed at baseline, pre-discharge (approximately 50 days following residential admission), and 1-, 2-, and 3-months post-residential-treatment discharge.
  Cognitive and Affective Mindfulness Scale (Feldman et al., 2007). Scores for this scale range from 10 to 40 with higher scores reflecting greater dispositional mindfulness (i.e., favorable outcomes). Scores for this measure will determine the changes across time (i.e., pre-post treatment and follow-up phases of study).
MBRP Treatment Adherence | Assessed for MBRP participants during residential treatment (~5 weeks)
  Number of MBRP sessions attended and self-report measures recording homework completion (e.g., frequency/duration of meditation practices).
Reward Probability | Assessed at baseline, pre-discharge (approximately 50 days following residential admission), and 1-, 2-, and 3-months post-residential-treatment discharge.
  Reward Probability Inventory (Carvalho et al., 2011). Scores for this scale range from 20 to 80 with higher scores reflecting greater perceived access to and engagement in rewarding and pleasurable activities (i.e., favorable outcomes). Scores for this measure will determine the changes across time (i.e., pre-post treatment and follow-up phases of study).
Post-Discharge Treatment Utilization | Assessed 1-, 2-, and 3-months post-residential-treatment discharge.
  Assessment of behavioral treatment services used during post-discharge follow-up assessment time-points.
Patient Reported Outcomes - Mental Health | Assessed at baseline, pre-discharge (approximately 50 days following residential admission), and 1-, 2-, and 3-months post-residential-treatment discharge.
  Assessed with the Patient-Reported Outcomes Measurement Information. System (Cella et al., 2010). Scores for this scale range from 4 to 20 with higher scores reflecting greater overall mental health (i.e., favorable outcomes). Scores for this measure will determine the changes across time (i.e., pre-post treatment and follow-up phases of study).

CONTACTS AND LOCATIONS:
Overall Officials: Michael J Gawrysiak, PhD, Principal Investigator — West Chester University of Pennsylvania
Locations (1):
- Gaudenzia, Inc. (West Chester House), West Chester, Pennsylvania, United States

IPD SHARING:
Plan to Share IPD: Yes
After all primary analyses and reports have been generated by the study PI to satisfy the aims of the research proposal, the PI will accept requests for components of the data to be available to other researchers for secondary analyses. When appropriate, the PI will share information necessary to foster productive collaborations.
Supporting Information: Study Protocol, SAP, ICF
Time Frame: When deemed appropriate by the study PI, data will be available after all primary research questions, statistical analyses, and publications have been completed.
Access Criteria: Submission of a formal request to the study PI indicating what specific information is requested and what the intentions are for use of this data.